CLINICAL TRIAL: NCT03866733
Title: Lecturer of Anesthesia, Intensive Care and Pain Management in Ain Shams University
Brief Title: Continuous Erector Spinea Block Versus Intravenous Analgesia in Coronary Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sanaa Farag Mahmoud Wasfy, lecturer of aneathesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R07l2019
Record Dates: First submitted 2019-03-03; First posted 2019-03-07 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Erector Spinea Block in Open Heart Surgery
Keywords: erector spinea block, open heart surgeries,analgesia
MeSH Terms: conditions — Agnosia | interventions — Narcotics; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Narcotics group (group N) (Active Comparator): intervention: injection of boluses of intra venous Narcotics (fentanyl) in the dose of (3-5 mcg/kg) during the surgery after induction of anesthesia. morphine 0.5mg/kg as rescue analgesia will be started upon arrival till 48 hours after surgery. NSAID every 12 hrs if there is no contraindication and iv acetaminophine igm/6hrs.
  Interventions: Drug: intravenous narcotics
- Erector spinea block group (group B) (Experimental): intervention: after induction our intervention will be the performance of ultrasound guided bilateral continous Erector spinea block with insertion of catheters then 15 ml of 0.25% bupivacaine will be injected in each of the catheters followed by a continuous infusion of 0.125% plain bupivacaine at the rate of 8 ml/h. morphine 0.5mg/kg as rescue analgesia will be started upon arrival till extubation and iv acetaminophine igm/6hrs.
  Interventions: Other: continous erector spinea block

INTERVENTIONS:
Other: continous erector spinea block — Ultrasound guided erector spinea block will be performed while the patient is in left lateral position ) the US probe will be placed in longitudinal parasagittal plane lateral to the T5 spinous process. An 18-gauge epidural needle will be inserted in-plane in a cranial-to-caudal direction until the tip is deep to erector spinae muscle. A 5 cm of epidural catheter will be threaded in cephalad direction. The same steps will be performed on the other side, after the negative aspiration for blood, bolus dose 15 ml of 0.25% bupivacaine will be injected in each of the catheters followed by a continuous infusion of 0.125% plain bupivacaine at the rate of 0.1 ml/kg/h.
  Arms: Erector spinea block group (group B)
Drug: intravenous narcotics — intervention: injection of boluses of intra venous Narcotic drugs (fentanyl) in the dose of (1-2mcg/kg) during the surgery after induction of anesthesia then fentanyl infusion through the postoperative first 24 hours postoperative till extubation then intravenous pethidine till 48 hours after surgery.
  Other Names: iv narcotics and NSAID
  Arms: Narcotics group (group N)

SUMMARY:
Adequate postoperative pain relief in patients in cardiac surgery is very essential. multimodal techniques for perioperative pain management post cardiac surgery include intravenous patient controlled analgesia, thoracic epidural and paravertebral blockade. Analgesia through thoracic epidural is the gold standard technique for post-sternotomy pain control but it has serious complications. ESP block is an easy technique compared to paravertebral block and less hazardous than thoracic epidural. Hence, this study will compare continuous bilateral erector spinae block guided by ultrasound with intravenous analgesia which is the standard method for pain management in cardiac surgery.

DETAILED DESCRIPTION:
Analgesia through thoracic epidural is the gold standard technique for post-sternotomy pain control. in spite of its serious complications such as epidural hematoma with or without paraplegia that enhanced by heparin administered during cardiac bypass surgery..

Paravertebral blockade is comparable to Thoracic epidural analgesia in cardiac surgery but it may cause complications such as vascular injuries and pneumothorax.

Erector spinae block is recently implemented technique for treatment and analgesia of thoracic neuropathic pain and post mastectomy syndrome. ESP block is an easy technique compared to paravertebral block and less hazardous than thoracic epidural.

This study will compare continuous bilateral erector spinae block guided by ultrasound versus intravenous analgesia for pain management in cardiac surgery Patients will be enrolled in the study will be divided into two groups In Group A: 20 patients will receive fentanyl after induction and intubation in the dose of ( 3-52mcg/kg ) according to the patients haemodynamic parameters and the decision of the anaesthesia team at skin incision, before starting Cardiopulmonary bypass and again after bypass and before sternal closure. Once the surgical procedure is ﬁnished, patients will be transferred to ICU. After ICU transfer acetaminophen 1 gm/6hrs will be given regularly and NSAID if there is no contraindication after extubation. morphine 0.5mg/kg as rescue analgesia will be started upon arrival till extubation.

In Group B: 20 patients will have bilateral ESP block will be done under general anaesthesia bolus dose 15 ml of 0.25% bupivacaine will be injected in each of the catheters followed by a continuous infusion of 0.125% plain bupivacaine at the rate of 8 ml/h starting in ICU for 48 h after extubation. patients will receive intraoperative boluses of fentanyl according to the patients' haemodynamic and the decision of the anaesthesia team at skin incision, before starting Cardiopulmonary bypass and again after bypass and before sternal closure. Once the surgical procedure is ﬁnished, patients will be transferred to ICU morphine 0.5mg/kg as rescue analgesia will be started upon arrival till extubation. Infusion rate will be titrated according to haemodynamics, pain assessment, and complications. After extubation acetaminophen 1gm/6hrs will be given regularly.

ELIGIBILITY:
Inclusion Criteria:

* elective cardiac surgery.
* age 18-65 years.
* patients with median sternotomy.
* body mass index <30kg.m2.
* left ventricular ejection fraction >50%.

Exclusion Criteria:

* signiﬁcant aortic stenosis.
* left main coronary artery disease.
* patient on anti-coagulants0
* pre-existing respiratory, neurological, or renal disease.
* CSF or blood tap during the procedure.
* failure to thread the catheter.
* anomalies of vertebral column.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
effectiveness of perioperative analgesia | 48 hours after surgery
  total dose of perioperative narcotics

SECONDARY OUTCOMES:
extubation time | 12 hours after end of surgery
  time passed between end of surgery and removal of endotracheal tube

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Sanaa Farag Mahmoud, Cairo, New Cairo
  - Ainshams hospitals, Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fibla JJ, Molins L, Mier JM, Sierra A, Vidal G. Comparative analysis of analgesic quality in the postoperative of thoracotomy: paravertebral block with bupivacaine 0.5% vs ropivacaine 0.2%. Eur J Cardiothorac Surg. 2008 Mar;33(3):430-4. doi: 10.1016/j.ejcts.2007.12.003. Epub 2008 Jan 16. PMID 18201893
- [Background] Raksamani K, Wongkornrat W, Siriboon P, Pantisawat N. Pain management after cardiac surgery: are we underestimating post sternotomy pain? J Med Assoc Thai. 2013 Jul;96(7):824-8. PMID 24319854
- [Background] Hansdottir V, Philip J, Olsen MF, Eduard C, Houltz E, Ricksten SE. Thoracic epidural versus intravenous patient-controlled analgesia after cardiac surgery: a randomized controlled trial on length of hospital stay and patient-perceived quality of recovery. Anesthesiology. 2006 Jan;104(1):142-51. doi: 10.1097/00000542-200601000-00020. PMID 16394700
- [Background] Dhole S, Mehta Y, Saxena H, Juneja R, Trehan N. Comparison of continuous thoracic epidural and paravertebral blocks for postoperative analgesia after minimally invasive direct coronary artery bypass surgery. J Cardiothorac Vasc Anesth. 2001 Jun;15(3):288-92. doi: 10.1053/jcan.2001.23271. PMID 11426357
- [Background] Canto M, Sanchez MJ, Casas MA, Bataller ML. Bilateral paravertebral blockade for conventional cardiac surgery. Anaesthesia. 2003 Apr;58(4):365-70. doi: 10.1046/j.1365-2044.2003.03082_2.x. PMID 12688271